CLINICAL TRIAL: NCT03800602
Title: Phase II Trial of Nivolumab and Metformin in Patients With Treatment Refractory MSS Metastatic Colorectal Cancer
Brief Title: Nivolumab and Metformin in Patients With Treatment Refractory MSS Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Olumide Gbolahan, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00106678; NCI-2018-02201 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4494-18 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Adenocarcinoma; Metastatic Microsatellite Stable Colorectal Carcinoma; Refractory Colorectal Carcinoma; Stage IV Colorectal Cancer; Stage IVA Colorectal Cancer; Stage IVB Colorectal Cancer; Stage IVC Colorectal Cancer; Colorectal Cancer Metastatic
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Metformin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, metformin) (Experimental): Patients receive metformin PO BID starting on day 1. After 14 days of metformin only period patients also receive nivolumab IV every 4 weeks starting on day 15. Courses repeat every 28 days for up to 2 years in the absence of disease progression, unacceptable toxicity or consent withdrawal.
  Interventions: Drug: Metformin; Biological: Nivolumab

INTERVENTIONS:
Drug: Metformin — Given PO
  Other Names: Glucophage; Glumetza; Fortamet
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies how well nivolumab and metformin work in treating patients with microsatellite stable (MSS) stage IV colorectal cancer that has not responded to previous treatment. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Metformin is an antidiabetic drug that and may reduce the risk of colorectal cancer development in patients. Giving nivolumab and metformin may work better in treating patients with refractory microsatellite metastatic colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of nivolumab and metformin combination on the overall response rate (ORR) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

SECONDARY OBJECTIVES:

I. To determine the effect of nivolumab and metformin combination on clinical outcomes, progression free survival and overall survival, and biochemical response (CEA).

II. To compare the effect of nivolumab and metformin combination on immune and metabolic biomarkers in the tumor microenvironment and systemic circulation (pre and post treatment paired biopsies required).

OUTLINE:

Patients receive metformin PO BID starting on day 1. After 14 days of metformin only period patients also receive nivolumab IV every 4 weeks starting on day 15. Courses repeat every 28 days for up to 2 years in the absence of disease progression, unacceptable toxicity or consent withdrawal

After completion of study treatment, patients are followed up at day 30 and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage IV colorectal adenocarcinoma with measurable disease
* Prior treatment with 5 Fluorouracil (or capecitabine), oxaliplatin and irinotecan containing chemotherapy (needs to be treated with anti-epidermal growth factor receptor (EGFR) agent if extended RAS wild type)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 (Karnofsky ≥ 70%)
* Life expectancy of greater than 3 months
* Absolute neutrophil count ≥ 1,500/µL
* Platelets ≥ 100,000/µL
* Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) OR creatinine clearance ≥ 60 mL/min/1.73 m² for patients with creatinine levels > 1.5 x ULN. Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin ≤ 1.5 x the upper limit of normal (ULN) OR direct bilirubin ≤ ULN for subjects with total bilirubin > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase[SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT] ≤ 2.5 x institutional upper limit of normal
* Serum albumin ≥ 2.5 mg/dl
* International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants. Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Patients with diabetes mellitus should be on a stable diabetic treatment regimen for at least 1 month prior to trial enrollment and keep a blood glucose level log at home for the first 4 weeks of the trial
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier

  * Note: Subjects with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Metformin use in the last 3 months
* Patients who are receiving any other investigational agents
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab and metformin
* Has a known history of active tuberculosis (TB) (Bacillus tuberculosis)
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has known substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Has received prior therapy with an anti-programmed death (PD)-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy.

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or myocardial infraction within 6 months of study entry, serious cardiac arrhythmia requiring medications, baseline corrected QT (QTc) > 450 msec or previous history of QT prolongation while taking other medications
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer; subjects with prior malignancies are eligible if the subject has been disease free for > 5 years
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2021-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olumide B. Gbolahan, MBBS, MSc, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

REFERENCES:
- [Derived] Akce M, Farran B, Switchenko JM, Rupji M, Kang S, Khalil L, Ruggieri-Joyce A, Olson B, Shaib WL, Wu C, Alese OB, Diab M, Lesinski GB, El-Rayes BF. Phase II trial of nivolumab and metformin in patients with treatment-refractory microsatellite stable metastatic colorectal cancer. J Immunother Cancer. 2023 Oct;11(10):e007235. doi: 10.1136/jitc-2023-007235. PMID 37852737

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Nivolumab, Metformin)
Started | 29
Completed | 24
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab, Metformin)
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 5
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [50 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Response will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1., and rate will be calculated as a proportion (responders/total patients).
Time Frame: Up to 1 year after study start
Population: 6 patients were replaced per protocol, and 18 patients had evaluable disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nivolumab, Metformin)
Number analyzed (Participants) | 18
Participants
  Stable Disease | 2
  Progressive Disease | 16

2. Secondary Outcome: Progression Free Survival (PFS)
Description: For progression free survival, progression or death from any cause will be defined as the event. Patients will be censored at time of last follow-up.
Time Frame: Assessed up to 2 years after study start
Population: 6 patients were replaced per protocol, and 18 patients had evaluable disease.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab, Metformin)
Number analyzed (Participants) | 18
months | 2.3 [1.7 to 2.3]

3. Secondary Outcome: Overall Survival (OS)
Description: For overall survival, death from any cause will be defined as the event. Patients will be censored at time of last follow-up.
Time Frame: Assessed up to 2 years after study start
Population: 6 patients were replaced per protocol, and 18 patients had evaluable disease.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nivolumab, Metformin)
Number analyzed (Participants) | 18
months | 5.2 [3.2 to 11.7]

4. Secondary Outcome: Biological Response: Carcinoembryonic Antigen (CEA)
Description: Tumor marker carcinoembryonic antigen (CEA) will be assessed.
Time Frame: Up to 1 year after study start
Population: This outcome was not analyzed because the data were not collected.
Arm/Group | Treatment (Nivolumab, Metformin)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued through the final assessment at Month 12.
Arm/Group | Treatment (Nivolumab, Metformin)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 18/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment (Nivolumab, Metformin) (N=18)
Diarrhea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 6
Abdominal Pain (General disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 5
Anemia (Blood and lymphatic system disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Fever (General disorders) | 3
Weight Loss (Metabolism and nutrition disorders) | 3
Abdominal Distension (Gastrointestinal disorders) | 2
Anxiety (Psychiatric disorders) | 2
Ast Increased (Blood and lymphatic system disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Lower Back Pain (Musculoskeletal and connective tissue disorders) | 2
Pelvic Pain (General disorders) | 2
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 2
Abdominal Cramps (Gastrointestinal disorders) | 1
Alk Phos Increased (Blood and lymphatic system disorders) | 1
B/L Le Edema (Vascular disorders) | 1
Bloating (Gastrointestinal disorders) | 1 (1)
Blood in Ostomy (Blood and lymphatic system disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1/9 (1)
Clostridioides Difficile Colitis (Gastrointestinal disorders) | 1
Decreased Appetite (General disorders) | 3
Dyphasia (General disorders) | 1 (1)
Elevated Ldh (Blood and lymphatic system disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Hyperbilirubinemia (General disorders) | 1
Hyperhidrosis (Night Sweats) (General disorders) | 1
Hypoalbuminemia (Blood and lymphatic system disorders) | 2
Hypokalemia (Blood and lymphatic system disorders) | 1
Left Hip Pain (Musculoskeletal and connective tissue disorders) | 1
Left Hydronephrosis (Renal and urinary disorders) | 1
Liver Failure (Endocrine disorders) | 1
Lle Dvt (Blood and lymphatic system disorders) | 1
Loss Of Bladder Control (Renal and urinary disorders) | 1
Loss Of Taste (General disorders) | 1
Lower Extremity Swelling (General disorders) | 1
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 1
Mouth Lesion (Skin and subcutaneous tissue disorders) | 1
Neck Pain (General disorders) | 1
Netropenia (General disorders) | 1
Pain At Biopsy Site (Skin and subcutaneous tissue disorders) | 1
Pain Lower Abdomen (Gastrointestinal disorders) | 1
Pulmonary Emoblism (Blood and lymphatic system disorders) | 1
Rash Underbreast (Skin and subcutaneous tissue disorders) | 1
Rectal Discharge (Renal and urinary disorders) | 1
Rectal Obstruction (Gastrointestinal disorders) | 1
Rectal Pain (Gastrointestinal disorders) | 1
Right Droopy Eye (Eye disorders) | 1
Right Internal Juglar Vein Thrombus (Injury, poisoning and procedural complications) | 1
Sepsis (Infections and infestations) | 1
Skin Itching (Skin and subcutaneous tissue disorders) | 1
Upper Back Pain (Musculoskeletal and connective tissue disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/02/NCT03800602/Prot_SAP_001.pdf
  • Informed Consent Form (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT03800602/ICF_000.pdf